CLINICAL TRIAL: NCT05707039
Title: Comparison of Open and Closed Chain Exercises on Pain Function and Balance in Athletes With Patellofemoral Pain Syndrome
Brief Title: Comparison of Open and Closed Chain Exercises in Athletes With Patellofemoral Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0406
Record Dates: First submitted 2023-01-22; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: PFPS, OCKE, CCKE
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open chain kinetic exercises (Experimental): In open chain exercises extremities are free to move and there is no weight bearing. Subjects performed group of exercises, 3sets of 10 repetitions for each exercise after warm-up and stretching exercises The open kinetic chain exercise program consisted of 1) maximal static quadriceps muscle contractions
  Interventions: Other: Open kinetic chain exercises
- Closed Chain Kinetic Exercises (Experimental): In closed kinetic chain exercises extremities are fixed and weight bearing is done. Subjects performed group of exercises, 3sets with 10 repetitions for each exercise after warm up and stretching exercises. The closed kinetic chain exercise program consisted of 1) seated leg presses, 2) one-third knee bends on one leg and on both legs, 3) stationary bicycling, 4) rowing-machine exercises, 5) step-up and step-down exercises. Each exercise in the closed kinetic chain protocol was performed dynamically with a 3-second rest between repetitions.
  Interventions: Other: Closed kinetic chain exercises

INTERVENTIONS:
Other: Open kinetic chain exercises — In open chain exercises extremities are free to move and there is no weight bearing.
  Arms: Open chain kinetic exercises
Other: Closed kinetic chain exercises — In closed kinetic chain exercises extremities are fixed and weight bearing is done.
  Arms: Closed Chain Kinetic Exercises

SUMMARY:
Patellofemoral pain syndrome (PFPS) is a common source of knee pain in the physically active population, predominantly in women. The incidence rate of PFPS among athletes is 25 percent, which is higher than that of general population. PFPS is caused by repetitive stress and aggravated in athletes by cycling and running. These symptoms are caused by structural or biomechanical changes of the joint, which becomes exacerbated by activities such as going up and down stairs, sit for a prolonged period, squatting or kneeling, resulting in increased compressive forces in the joint patellofemoral. It is characterized by defused pain in front of knee. Other signs also present are the patellar crepitus, swelling, and joint blockage despite being deemed a multifactorial condition with no single cure, PFPS is commonly attributed to muscular dysfunction, for which conservative rehabilitation is the treatment of choice. Historically, PFPS has been linked to impairments of the quadriceps muscle.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial will be conducted in Pakistan sports board Lahore, Model town Sports Club Lahore and Sheikh Zaid Hospital, Lahore. Sample size will be taken to evaluate the effects of open chain exercise and closed chain exercise among athletes with an age group of 18 - 40 years. Non probability convenient sampling technique would be used. Players having an experience of at least 8 months would be a part of study experiencing recurrent knee pain. Participants will be randomly assigned to 2 groups. Group A will include participants who will receive open kinetic chain exercises 3sets of 10 repetitions for each exercise along with the general training. Group B will include the participants who will receive closed kinetic chain exercises 3sets of 10 repetitions for each exercise along with general training.3sessions per week will be given for 6weeks.The subjects will be assessed for pain, function and balance at baseline and after 6weeks of treatment. After collecting data from defined settingit will be entered and analyzed using statistical package for social sciences (SPSS) for Windows software, version 25.

ELIGIBILITY:
Inclusion Criteria:

* Adult athletes with age 18 to 30 years
* Anterior Knee pain
* An insidious onset of symptoms not related to trauma.
* Pain with compression of patella.
* Pain on palpation of patellar facets.
* Experienced players (who are in practice from last 8 months or a year).

Exclusion Criteria:

* Symptoms present less than 1 month.
* Intra-articular knee pathologies like O.A, R.A etc
* History of knee surgery within last year.
* History of traumatic injuries like patellar dislocations or subluxation
* Any other lower extremity injuries.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
NPRS | 6 weeks
  Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale.
LEFS | 6 week
  Lower Extremity Functional Scale (LEFS) is to measure "patients' initial function, ongoing progress, and outcome" for a wide range of lower-extremity conditions.
Y balance test | 6 weeks
  Y Balance test is a dynamic test required for proprioception along with strength and flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asrar Yousaf, mphil, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No